CLINICAL TRIAL: NCT05336669
Title: Coagulation Profile in Patients Undergoing Coronary Intervention Measured With Activated Clotting Time, Global Thrombosis Test and Platelet Inhibition VerifyNow P2Y12 Test
Brief Title: Coagulation Profile in Patients Undergoing Coronary Angiography and Percutaneous Coronary Intervention
Acronym: GlobalACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: 69/VII/Budaj/2021
Record Dates: First submitted 2021-09-24; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-09

CONDITIONS: Chronic Coronary Insufficiency; Smoking
Keywords: coronary angiography; activated clotting time; platelet inhibition
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2ml sample of full blood from each patient at baseline 4ml sample of plasma from each patient at each timepoint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-smoking: Non-smoking patients undergoing coronary angiography or percutaneous coronary intervention
- Smoking: Smoking patients undergoing coronary angiography or percutaneous coronary intervention

SUMMARY:
The activated clotting time (ACT), global thrombosis test (GTT-3), platelet inhibition P2Y12 (VerifyNow) test and serum coagulation factors will be measured in patients undergoing coronary angiography (CA) and percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The activated clotting time (ACT), global thrombosis test (GTT-3) and platelet inhibition P2Y12 (VerifyNow) test and serum coagulation factors will be measured in patients undergoing coronary angiography (CA) and percutaneous coronary intervention (PCI) - 20 smoking and 20 non-smoking.The measurements will take place: before coronary angiography (CA), 10 minutes after unfractionated heparin (HNF), 2h after CA, 6h after CA, 30 days after CA

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled do CA >18 years old

Exclusion Criteria:

* pregnancy
* previous treatment with P2Y12 inhibitors, novel oral anticoagulants (NOAC) or warfarin acenocoumarol in last 24 hours

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients, 20 smoking at least 10 cigarettes a day, 20 patients non-smoking (<1 cigarette in last 30 days)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
ACT change | Baseline ACT , 10 minutes ACT, 2 hours ACT, 6 hours ACT, 30 days ACT
  Activated Clotting Time
GTT-3 change | Baseline GTT-3, 10 minutes GTT-3, 2 hours GTT-3, 6 hours GTT-3, 30 days ACT
  Global Thrombosis Test
VerifyNow change | Baseline VerifyNow, 10 minutes VerifyNow, 2 hours VerifyNow, 6 hours VerifyNow, 30 days ACT
  Platelet inhibition P2Y12 test

CONTACTS AND LOCATIONS:
Overall Officials: Bogumił Ramotowski, Principal Investigator — Centre of Postgraduate Medical Education

REFERENCES:
- [Derived] Ramotowski B, Lewandowski P, Slomski T, Maciejewski P, Budaj A. Platelet reactivity and activated clotting time predict hemorrhagic site complications in patients with chronic coronary syndromes undergoing percutaneous coronary interventions. Coron Artery Dis. 2024 Jun 1;35(4):292-298. doi: 10.1097/MCA.0000000000001336. Epub 2024 Jan 22. PMID 38241058